CLINICAL TRIAL: NCT02126657
Title: Phase 2 Study of the The Efficacy and Safety of a Single 70% Glycolic Acid Peel With Vitamin C for the Treatment of Acne Scars
Brief Title: The Efficacy and Safety of a Single 70% Glycolic Acid Peel With Vitamin C for the Treatment of Acne Scars
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013/01230
Record Dates: First submitted 2014-04-28; First posted 2014-04-30 (Estimated); Last update posted 2014-04-30 (Estimated); Status verified 2014-04

CONDITIONS: Acne Scars
Keywords: Acne scars; 70% Glycolic acid peel
MeSH Terms: interventions — glycolic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Other): Single arm study - pre and post peel assessment
  Interventions: Drug: 70% glycolic acid

INTERVENTIONS:
Drug: 70% glycolic acid

SUMMARY:
Our study involves the evaluation of a high potency chemical peel in its efficacy and safety profile for the treatment of acne scars. This chemical peel regime is a high potency peel of 70% glycolic acid combined with vitamin C that is purported to provide a good balance between yielding results and patient safety. We aim to evaluate its efficacy and safety profile of a single application. The study design is based on a single group that compares pre- vs post-intervention. 10 patients with atrophic acne scars of skin type I-IV will be recruited. Potential benefits include improvement of post acne scars with a short downtime and risks include post peel hyper pigmentation and scarring. We believe that this treatment will be highly beneficial to patients with post acne scarring.

This chemical peel regime has good efficacy and safety profile for the treatment of acne scars.

DETAILED DESCRIPTION:
Primary endpoints:

1. ECCA (échelle d'évaluation clinique des cicatrices d'acné) grading scale for quantitative grading of acne scars. Two blinded evaluators compare and rate the photograph using ECCA score.
2. Patient Assessment Based on 1 to 10 point scale; 1- nil acne scars and 10- severe acne scar

Secondary endpoints:

1. Postacne hyperpigmentation index (PAHPI)

   -Each of these 3 variables --size, intensity, and number of lesions is weighted and the summation of the weighted variables gives the total PAHPI score, ranging 6 to 22.
2. Safety Assessment (This is an ordinal scale) i. Score of redness ii. Score of swelling iii. Score of oozing/crusting iv. Post peel hyperpigmentation v. Post peel scarring vi. Assessment based on patient and doctor global assessment (global assessment from 1 - 10)

ELIGIBILITY:
Inclusion Criteria:

1. Atrophic scars
2. Skin type I to IV

Exclusion Criteria:

1. Pregnancy, breastfeeding
2. Active dermatitis (on the face), rosacea, allergic rhinitis, active herpes simplex
3. Known hypersensitivity
4. Previous keloids
5. Laser ablative procedures within the last month
6. Chemical peels within the last 6 months
7. Used oral retinoids in the past 6 months
8. Used topical retinoids in the past one week
9. Used scrub, AHA, skin irritant for the past 24h
10. Presence of facial warts or fungal infections
11. Photoallergies
12. Prior poor reaction to a chemical peel
13. Radiotherapy
14. Skin type V and VI
15. Patients with predominantly ice pick and boxcar scars

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-05; Primary Completion 2014-11 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Efficacy Assessment | 3 months
  1. ECCA (échelle d'évaluation clinique des cicatrices d'acné) grading scale for quantitative grading of acne scars
     * V-shaped atrophic scars with diameter <2 mm: 15
     * U-shaped atrophic scars with a diameter of 2-4 mm: 20
     * M-shaped atrophic scars with diameter >4 mm: 25
     * Superficial elastolysis: 30
     * Hypertrophic scars with a <2-year duration: 40
     * Hypertrophic scars of >2-year duration: 50 A semi-quantitative scoring of number of each scar will be performed
     * No scars: 0
     * Less than five scars: 1
     * Between five and 20 scars: 2
     * More than 20 scars: 3
  2. Patient Assessment Based on 1 to 10 point scale; 1- nil acne scars and 10- severe acne scar
  Secondary endpoints
  1) Postacne hyperpigmentation index (PAHPI)
Safety Assessment | 3 months
  ) Safety Assessment (This is also an ordinal scale) i. Score of redness ii. Score of swelling iii. Score of oozing/crusting iv. Post peel hyperpigmentation v. Post peel scarring

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore